CLINICAL TRIAL: NCT01108601
Title: Transtympanic Administration of Lactate: An Innovative Otoprotection for Patients Receiving Cisplatin or Carboplatin Chemotherapy
Brief Title: Transtympanic Ringer's Lactate for the Prevention of Cisplatin Ototoxicity
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Dr. Sam Daniel, McGill University Health Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GEN-07-033
Record Dates: First submitted 2010-04-01; First posted 2010-04-22 (Estimated); Last update posted 2010-04-22 (Estimated); Status verified 2010-04

CONDITIONS: Hearing Loss
Keywords: Ringer's; lactate; cisplatin; ototoxicity; hearing loss
MeSH Terms: conditions — Hearing Loss; Ototoxicity | interventions — Ringer's Lactate; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ringer's Lactate (Other): Each patient will act as their own control with one ear receiving treatment, and the contralateral ear acting as control.
  Interventions: Drug: Ringer's Lactate (0.03% Ciprofloxacin)

INTERVENTIONS:
Drug: Ringer's Lactate (0.03% Ciprofloxacin) — For each patient, only one ear will receive the Ringer's Lactate solution. The other ear will act as a control. To ensure adequate delivery of the solution to the middle ear, a small pressure equalizing tube will be inserted under local anesthesia before commencement of chemotherapy treatment. The patient will be instructed to administer four drops of RL solution to the experimental ear twice a day during their chemotherapy treatment.

SUMMARY:
Cisplatin and carboplatin induce ototoxicity manifested as sensorineural hearing loss, tinnitus, and/or vestibular disturbances. Ototoxicity is induced via damage to inner ear structures by reactive oxygen species. Previous animal studies demonstrated that transtympanic injection of Ringer's Lactate (RL) provided near complete otoprotective effect against cisplatin. The purpose of this study is to determine if transtympanic administration of Ringer's Lactate via a pressure equalising (PE) tube in patients undergoing platinum based chemotherapy treatment will prevent tinnitus, vestibular dysfunction and hearing loss especially at high frequencies. Pre- and post- chemotherapy treatment audiometry will be measured and statistically analysed for significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 14
* Patients undergoing platinum based chemotherapy
* Patients who agree to participate in the study

Exclusion Criteria:

* Patients unable to provide consent
* Patients with head and neck cancer
* Patients undergoing radiation of the head and neck
* Patients who develop a tympanic perforation
* Patients with persistent otorrhea

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Audiogram | Before and after chemotherapy treatment
  Pre-, mid-(if available) and post-chemotherapy treatment audiograms will be compared to determine changes in hearing from baseline and between ears. Hearing will also be assessed every six months after chemotherapy treatment for up to four years to determine possible long-term effects.

SECONDARY OUTCOMES:
Otoacoustic Emissions | Before and after chemotherapy treatment
  Distortion Product Otoacoustic Emissions will also be measured before and after chemotherapy treatment and compared to determine significance.

CONTACTS AND LOCATIONS:
Overall Officials: Sam J Daniel, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Choe WT, Chinosornvatana N, Chang KW. Prevention of cisplatin ototoxicity using transtympanic N-acetylcysteine and lactate. Otol Neurotol. 2004 Nov;25(6):910-5. doi: 10.1097/00129492-200411000-00009. PMID 15547419
- See also: Protection From Cisplatin Ototoxicity by Lactated Ringers — http://clinicaltrials.gov/ct2/show/NCT00584155?term=ringer%27s+lactate&rank=2